CLINICAL TRIAL: NCT07096986
Title: Impact of Dapagliflozin for the Regulation of Immunological Activity in Membranous
Brief Title: Impact of Dapagliflozin for the Regulation of Immunological Activity in Membranous Nephropathy
Acronym: FORXIGEM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-AOIP-06
Record Dates: First submitted 2025-07-07; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FORXIGA (Experimental)
  Interventions: Drug: Forxiga

INTERVENTIONS:
Drug: Forxiga — dapagliflozin treatment at a dose of 10 mg per os daily for 6 months

SUMMARY:
WHY IS THIS RESEARCH BEING CONDUCTED? Membranous glomerulonephritis (MN) is an autoimmune disease that affects the kidneys through autoantibodies, meaning that antibodies produced by your body attack your own kidney cells. The appearance of these autoantibodies can be explained in part by a disruption in the immune response. Patients with this disease are treated with immunosuppressive drugs such as rituximab. The aim of this treatment is to reduce the production of all antibodies, including those responsible for the disease. Despite this treatment, some patients may experience a relapse of the disease. These relapses can be complicated by infections, blood clots in the blood vessels, and, in the long term, can lead to kidney failure and an increased cardiovascular risk. Relapses can also have an impact on patients' social and professional lives.

Dapagliflozin is a diuretic medication, which means that it is used to increase urine production and eliminate excess salt and water from the body to reduce edema (swelling). It is currently prescribed and authorized for patients with type 2 diabetes, heart failure and chronic kidney disease. This treatment has been shown to reduce the amount of proteins in the urine and protect the kidneys and cardiovascular system in patients with chronic kidney disease. A study has also shown that dapagliflozin may have an effect on the immune response.

WHAT DOES IT INVOLVE? The aim of our study will be to evaluate the efficacy of dapagliflozin in reducing disease autoantibodies and preventing relapses.

This research will be conducted at the Nice University Hospital and the Nîmes University Hospital. We expect to 20 patients to be recruited with an anti-PLA2R1 positive MN.

Participation in the study will last 6 months. The research is funded by Nice University Hospital. WHAT IS THE TREATMENT BEING STUDIED? It is dapagliflozin, a drug that is increasingly used routinely in patients with nephrotic syndrome (including MN) for its ability to reduce protein in the urine. Its effect on the immune system in MN has not yet been studied

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years old and < 85 years old;
* Membranous Nephropathy associated with anti-PLA2R1 autoantibodies;
* Urine Protein Creatinine Ratio (UPCR) between 0.5 g/g and 3.5 g/g;
* Immunological relapse defined by an increase in anti-PLA2R1 antibody concentration > 14 RU/mL after a phase of anti-PLA2R1 antibody negativation, (i.e. immunological remission) and complete or partial clinical remission;
* Antiproteinuric treatment at maximal and stable dose. According to KDIGO 2024 guidelines on management of glomerular diseases and the French recommendations (PNDS GEM 2022), symptomatic treatment of membranous nephropathy should include: (i) a low sodium diet, (ii) a diuretic and (iii) an angiotensin-converting enzyme inhibitor or an angiotensin 2 receptor blocker at maximal tolerated dose (i.e., absence of orthostatic hypotension and no increase in serum creatinine >30%).

Exclusion Criteria:

* Immunosuppressive treatment for MN in the 6 months prior to the selection visit;
* Secondary MN (associated with cancer, infectious disease, autoimmune or iatrogenic disease);
* Active nephrotic syndrome defined according to KDIGO guidelines as proteinuria > 3.5 g/day (or 3.5 g/g in a urine sample) and albumin < 30 g/L;
* No previous history of immunological remission (anti-PLA2R1 antibodies < 14 RU/mL in ELISA or negative indirect immunofluorescence) or clinical remission (partial or complete);
* Galactose intolerance, total lactase deficiency or glucose-galactose malabsorption disorders
* Patients at risk for ketoacidosis including patients with a low reserve of functional beta cells (e.g. patients with type 2 diabetes with low C-peptide or latent autoimmune diabetes mellitus or patients with a history of pancreatitis or patients who are receiving insulin treatment), patients with conditions leading to reduced food intake or severe dehydration, patients with low insulin reserve, and patients with increased insulin requirements due to acute medical illness, surgery or excessive alcohol consumption;
* Type 1 diabetes;
* Pregnancy or breastfeeding;
* Estimated CKD-EPI Glomerular Filtration Rate (eGFR) < 25 ml/min/1.73m2;
* Severe liver failure (Child-Pugh stage C);
* NYHA functional class IV heart failure;
* Patients already currently receiving dapagliflozin or another SGLT2 inhibitor for another condition;
* Repeated urinary tract infections;
* Hypersensitivity to the active substance or excipients.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To measure immunological activity (anti-PLA2R1 antibody concentration) in anti-PLA2R1 antibodies positive MN patients undergoing an immunological relapse, before and after 6 months of dapagliflozin treatment. | 6 months
  Change in anti-PLA2R1 antibody titer (ELISA titer in RU/mL) from baseline to 6 months after dapagliflozin treatment compared with pretreatment antibody titer.

SECONDARY OUTCOMES:
To measure the change in proteinuria over the course of the study in anti-PLA2R1 antibodies positive MN patients undergoing an immunological relapse | 6 months
  Change in proteinuria (in g/g) from baseline to 6 months after dapagliflozin treatment (under stable antiproteinuric treatment)
To measure the change in serum albumin levels over the course of the study in anti-PLA2R1 antibodies positive MN patients undergoing an immunological relapse | 6 months
  Change in albumin levels (in g/L) from baseline to 6 months after dapagliflozin treatment (under stable antiproteinuric treatment)
To measure the change in glomerular filtration rate over the course of the study in anti- PLA2R1 antibodies positive MN patients undergoing an immunological relapse | 6 months
  Change in glomerular filtration rate (in ml/min/1.73m2) from baseline to 6 months after dapagliflozin treatment (under stable antiproteinuric treatment)
To measure the occurrence of clinical relapses over the course of the study in anti-PLA2R1 antibodies positive MN patients undergoing an immunological relapse | 6 months
  Need for Rituximab treatment for clinical relapse (according to KDIGO 2021 guidelines and French 2022 guidelines)
To measure the production of Th17, Th2 and Treg pathway cytokines in anti-PLA2R1 antibodies positive MN patients undergoing an immunological relapse, before and after 6 months of dapagliflozin treatment | 6 months
  Change in cytokine profile from baseline to 6 months after dapagliflozin treatment
To assess the dapagliflozin treatment's safety in MN patients | 6 months
  Appearance of side effects
To assess the dapagliflozin treatment's safety in MN patients | 6 months
  Appearance of biological disorder

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
not scheduled